CLINICAL TRIAL: NCT02492425
Title: Evaluating the Adherence to Guidelines' Empirical Antibiotic Recommendations and Outcome of Patients Admitted to a Hospital Ward With a Diagnosis of Community-acquired Pneumonia
Brief Title: A Registry Study on Hospitalized Patients With Community-acquired Pneumonia in Real-life of China
Acronym: CAP-China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Bin Cao, MD, Capital Medical University
Other Study IDs: NCT20150401
Record Dates: First submitted 2015-03-16; First posted 2015-07-08 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Community Acquired Pneumonia
Keywords: Community Acquired Pneumonia; Healthcare Associated Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia; Healthcare-Associated Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the disease burden of hospitalized patients with CAP and HCAP in real life of China

DETAILED DESCRIPTION:
In China, the data about current management of patients hospitalized with community acquired pneumonia (CAP) in the real-life setting is not available,type of pneumonia, selection of initial antibiotic, time to clinical stability, antibiotic choice anf modification,clinical outcomes and costs remain unclear.

In this study, we will collect comprehensive information on CAP and healthcare associated pneumonia (HCAP) management patterns to evaluate the disease burden of hospitalized patients with CAP and HCAP in real life of China .to analyze microbiological characteristics,clinical manifestations,antibiotic regimens ,adherences to guidelines and effect on outcome in different groups of patients with CAP (> and = 65 years, different comorbidities ,risk factors) ,to investigate microbiological characteristics,clinical manifestations,antibiotic regimens ,adherences to guidelines and effect on outcome in different groups of disease severity with CAP ,to provide the difference on microbiological characteristics,clinical manifestations,antibiotic regimens ,and outcome between patients with CAP and HCAP ,to understand the current situation of antibiotic regimen ,to evaluate influence of different antibiotic regimens on prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients > or = 14 years of age
* Patient meets the criteria of community acquired pneumonia
* Patient meets the criteria of healthcare-associated pneumonia
* Informed consent to participate in the study is provided

Exclusion Criteria:

* Patients participating in a clinical trial or other intervention studies
* Patients <14 years of age
* Patient meets the criteria of hospital acquired pneumonia
* Known active tuberculosis or current treatment for tuberculosis
* Non-infectious pulmonary diseases （e.g. pulmonary embolism, pulmonary edema, pulmonary vasculitis, interstitial pneumonia）
* HIV positive

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 3000 patients with community acquired pneumonia who meet the below inclusion/ exclusion criteria will be recruited in China
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
initial antibiotic treatment failure rate | 72 hours
  a change in antibiotic therapy due to worsening signs or symptoms of infection or lack of clinical improvement after first dose use of antibiotics to 72h
in-hospital clinical failure rate | Time from date of admission to discharge up to 1 week
  1)a change in antibiotic therapy due to worsening signs or symptoms of infection or lack of clinical improvement, 2) in-hospital mortality, 3) recurrence, defined as signs or symptoms of infection after completion of therapy requiring re-initiation of antibiotics
30-day post-discharge clinical failure rate | discharge up to 5 weeks
  rate of re-hospitalization due to pulmonary infection and death during the follow-up period at 30 days post-discharge from hospital

SECONDARY OUTCOMES:
Duration of intravenous antimicrobial therapy | 2 weeks
  Time from the first dose of intravenous antibiotics to date of stop of intravenous antibiotics ,participants will be followed for the duration of hospital stay
Duration of oral antimicrobial therapy | 2 weeks
  Time from date of administration of first antibiotic to date of discontinuation of last antibiotic
Duration of antimicrobial therapy | 6 weeks
  Time from date of administration of first antibiotic to date of discontinuation of last antibiotic (or to date of censoring, whichever comes first) upto a maximum of 30 days post-discharge from hospital post discharge from hospital
Days of each antimicrobial therapy | 6 weeks
  Time from date of first administration on admission to hospital to date of discontinuation (or to date of censoring, whichever comes first) upto a maximum of 30 days post-discharge follow-up for each antibiotic
Hospital length of stay | 2 weeks
  Patients will be asked about hospitalization, date, Patients will be asked about hospitalization, date, participants will be asked about the time of admission and discharge

CONTACTS AND LOCATIONS:
Overall Officials: Bin Cao, MD, Study Chair — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, China

REFERENCES:
- [Result] Yang SQ, Qu JX, Wang C, Yu XM, Liu YM, Cao B. Influenza pneumonia among adolescents and adults: a concurrent comparison between influenza A (H1N1) pdm09 and A (H3N2) in the post-pandemic period. Clin Respir J. 2014 Apr;8(2):185-91. doi: 10.1111/crj.12056. Epub 2013 Nov 26. PMID 24106842
- [Result] Cao B, Huang GH, Pu ZH, Qu JX, Yu XM, Zhu Z, Dong JP, Gao Y, Zhang YX, Li XH, Liu JH, Wang H, Xu Q, Li H, Xu W, Wang C. Emergence of community-acquired adenovirus type 55 as a cause of community-onset pneumonia. Chest. 2014 Jan;145(1):79-86. doi: 10.1378/chest.13-1186. PMID 24551881
- [Result] Qu J, Gu L, Wu J, Dong J, Pu Z, Gao Y, Hu M, Zhang Y, Gao F, Cao B, Wang C; Beijing Network for Adult Community-Acquired Pneumonia (BNACAP). Accuracy of IgM antibody testing, FQ-PCR and culture in laboratory diagnosis of acute infection by Mycoplasma pneumoniae in adults and adolescents with community-acquired pneumonia. BMC Infect Dis. 2013 Apr 11;13:172. doi: 10.1186/1471-2334-13-172. PMID 23578215
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=Influenza+pneumonia+among+adolescents+and+adults%3A+a+concurrent+comparison+between+influenza+A+(H1N1)+pdm09+and+A+(H3N2)+in+the+post-pandemic+period.
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=Emergence+of+community-acquired+adenovirus+type+55+as+a+cause+of+community-onset+pneumonia
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=Accuracy+of+IgM+antibody+testing%2C+FQ-PCR+and+culture+in+laboratory+diagnosis+of+acute+infection+by+Mycoplasma+pneumoniae+in+adults+and+adolescents+with+community-acquired+pneumonia.